CLINICAL TRIAL: NCT03923673
Title: TtP: Minimally Invasive Pericardiotomy as a New Treatment for Heart Failure (Transform the Practice)
Brief Title: Minimally Invasive Pericardiotomy as a New Treatment for Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-010106
Record Dates: First submitted 2019-04-16; First posted 2019-04-22 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Pericardiectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with Heart Failure with Preserved Ejection Fraction (Experimental): Subjects with Heart Failure with Preserved Ejection Fraction (HFpEF) will receive a minimally invasive treatment called a pericardiotomy.
  Interventions: Procedure: Pericardiotomy

INTERVENTIONS:
Procedure: Pericardiotomy — The minimally invasive procedure that creates a small opening in the sac that surrounds the heart.

SUMMARY:
Researchers are studying the safety and efficacy of a minimally invasive treatment called a pericardiotomy, which creates a small opening in the sac that surrounds the heart. Researchers will test the short and long term effects of this procedure by monitoring subjects heart function and symptoms.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 30 years
* Symptoms of severe dyspnea (III-IV) without evidence of a non-cardiac or ischemic explanation for dyspnea
* EF of > or = 50% determined on most recent imaging study within the preceding 5 years, with no change in clinical status suggesting potential for deterioration in systolic function
* One of the following:

  * Previous hospitalization for HF with radiographic evidence (pulmonary venous hypertension, vascular congestion, interstitial edema, pleural effusion) of pulmonary congestion or
  * Catheterization documented elevated filling pressures at rest (PCWP ≥15 or LVEDP ≥18) or with exercise (PCWP ≥25) or
  * Elevated NT-proBNP (>400 pg/ml) or BNP(>200 pg/ml) or
  * Echo evidence of diastolic dysfunction/elevated filling pressures manifest by medial E/e' ratio≥15 and/or left atrial enlargement and chronic treatment with a diuretic for signs or symptoms of heart failure
* Heart failure is primary factor limiting activity as indicated by answering # 2 to the following question: My ability to be active is most limited by:

  * Joint, foot, leg, hip or back pain
  * Shortness of breath and/or fatigue and/or chest pain
  * Unsteadiness or dizziness
  * Lifestyle, weather, or I just don't like to be active
  * Ambulatory (not wheelchair / scooter dependent)

Exclusion Criteria

* Recent (< 1 month) hospitalization for heart failure
* Left or right ventricular dilatation noted on cardiac imaging study prior to enrollment (either echocardiography or MRI).
* Any hemoglobin (Hgb) < 8.0 g/dl within 30 days prior to randomization
* Any GFR < 20 ml/min/1.73 m2 within 30 days prior to randomization
* Significant alternative cause of dyspnea such as severe chronic obstructive pulmonary disease that is a primary contributor to symptoms in the opinion of the investigator
* Ischemia thought to contribute to dyspnea in the opinion of the investigator
* Acute coronary syndrome within 3 months defined by electrocardiographic (ECG) changes and biomarkers of myocardial necrosis (e.g., troponin) in an appropriate clinical setting (chest discomfort or anginal equivalent)
* PCI, coronary artery bypass grafting, or new biventricular pacing within past 3 months
* Obstructive hypertrophic cardiomyopathy
* Known infiltrative cardiomyopathy (amyloid)
* Pericardial disease (constriction, pericarditis, tamponade)
* Active myocarditis
* Complex congenital heart disease
* Active collagen vascular disease
* Significant valvular heart disease (greater than mild stenosis or greater than moderate regurgitant lesions)
* Acute or chronic severe liver disease as evidenced by any of the following: encephalopathy, variceal bleeding, INR > 1.7 in the absence of anticoagulation treatment
* Terminal illness (other than HF) with expected survival of less than 1 year
* Enrollment or planned enrollment in another therapeutic clinical trial in next 3 months.
* Inability to comply with planned study procedures
* Pregnancy or breastfeeding mothers

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events | 6 months
  The number of major cardiac and cerebrovascular events reported.
Change in left ventricular filling pressures during volume loading | baseline, 6 months
  The number of subjects to demonstrate an increase in pulmonary capillary wedge pressure in response to volume loading after pericardiotomy vs. prior to pericardiotomy.

SECONDARY OUTCOMES:
Change in Quality of Life | baseline, 6 months
  Measured using Kansas City Cardiomyopathy Questionnaire (KCCQ)
Change in exercise capacity | baseline, 6 months
  Measured by Cardiopulmonary Exercise Testing

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials